CLINICAL TRIAL: NCT02115204
Title: Adjuvant Chemotherapy of Breast Cancer: Sequential Chemotherapy vs. Standard Therapy. Prospective Randomised Comparison of 4 x Epirubicin and Cyclophosphamide (EC) --> 4 x Docetaxel (Doc) vs. 6 x CMF / CEF in Patients With 1 to 3 Positive Lymph Nodes
Brief Title: 4 x Epirubicin, Cyclophosphamide, Followed by 4 x Docetaxel Versus 6 x CMF / 6 x CEF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: West German Study Group (Other)
Collaborators: AGO Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC-Doc
Record Dates: First submitted 2014-04-08; First posted 2014-04-15 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Docetaxel; Methotrexate; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EC-Doc (Experimental): 4 cycles epirubicin + docetaxel (90/600) i.v., q = 3 weeks, followed by 4 cycles docetaxel (100) i.v., q = 3 weeks
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- CMF/CEF (Active Comparator): 6 cycles cyclophosphamide, methotrexate, 5-fluorouracil (CMF) (600/40/600) i.v., day 1 + 8, q = 4 weeks or 6 cycles cyclophosphamide, epirubicin, 5-fluorouracil (CEF) (500/100/500) i.v., day 1, q = 3 weeks
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Methotrexate; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: Epirubicin
Drug: Cyclophosphamide
Drug: Docetaxel
  Arms: EC-Doc
Drug: Methotrexate
  Arms: CMF/CEF
Drug: 5-fluorouracil
  Arms: CMF/CEF

SUMMARY:
Taxane-based adjuvant chemotherapy is standard in node-positive (N+) early breast cancer (BC). The magnitude of benefit in intermediate-risk N+ early BC is still unclear. West German Study Group and "Arbeitsgemeinschaft Gynäkologische Onkologie" (WSG-AGO) EC-Doc is a large trial evaluating modern sequential taxane-based chemotherapy in the subgroup with 1-3 involved lymph nodes (LN).

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Age 18-65 years
* Eastern Cooperative Oncology Group (ECOG) status < 2
* Surgery: R0-resection and >= 10 removed axillary lymph nodes
* M0 by chest x-ray, bone scintigraphy and liver sonography

Exclusion Criteria:

* Polyneuropathy
* Creatinin (serum) > 1,4 mg/dl; Bilirubin (serum) > 2,0 mg/dl
* Cardia dysfunction, ejection fraction < lower normal value of each institution
* Hematopoeitic insufficiency: leucocytes < 3,5 G/l, thrombocytes < 100 G/l
* second malignant neoplasia, except curatively treated basalioma of the skin
* Surgery before more the six weeks (42 days)
* Concurrent pregnancy; patients of childbearing potential must implement a highly effective (less than 1% failure rate) non-hormonal contraceptive measures during the study treatment
* Breast feeding woman
* Sequential breast cancer
* Reasons indicating risk of poor compliance
* Patients not able to consent

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2011 (Actual)
Dates: Start 2000-06; Primary Completion 2005-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Comparison of event-free survival | 60 months after end of treatment

SECONDARY OUTCOMES:
Comparison of overall survival | 60 months after end of treatment
Comparison of toxicity (measured as number of adverse events) | 60 months after end of treatment
Comparison of quality of life | 60 months after end of treatment
Comparison of cost effectiveness across the applied regimens in relation to event-free survival | 60 months after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Nitz, Prof. Dr., Principal Investigator — Ev. Hospital Bethesda, Moenchengladbach
Locations (1):
- Ev. Hospital Bethesda, Mönchengladbach, Germany

REFERENCES:
- [Result] Nitz U, Gluz O, Huober J, Kreipe HH, Kates RE, Hartmann A, Erber R, Moustafa Z, Scholz M, Lisboa B, Mohrmann S, Mobus V, Augustin D, Hoffmann G, Weiss E, Bohmer S, Kreienberg R, Du Bois A, Sattler D, Thomssen C, Kiechle M, Janicke F, Wallwiener D, Harbeck N, Kuhn W. Final analysis of the prospective WSG-AGO EC-Doc versus FEC phase III trial in intermediate-risk (pN1) early breast cancer: efficacy and predictive value of Ki67 expression. Ann Oncol. 2014 Aug;25(8):1551-7. doi: 10.1093/annonc/mdu186. Epub 2014 May 14. PMID 24827128
- [Result] Erber R, Gluz O, Brunner N, Kreipe HH, Pelz E, Kates R, Bartels A, Huober J, Mohrmann S, Moustafa Z, Liedtke C, Mobus V, Augustin D, Thomssen C, Janicke F, Kiechle M, Kuhn W, Nitz U, Harbeck N, Hartmann A. Predictive role of HER2/neu, topoisomerase-II-alpha, and tissue inhibitor of metalloproteinases (TIMP-1) for response to adjuvant taxane-based chemotherapy in patients with intermediate-risk breast cancer: results from the WSG-AGO EC-Doc trial. Breast Cancer Res Treat. 2015 Apr;150(2):279-88. doi: 10.1007/s10549-015-3310-x. Epub 2015 Feb 28. PMID 25721604
- [Derived] Gluz O, Liedtke C, Huober J, Peyro-Saint-Paul H, Kates RE, Kreipe HH, Hartmann A, Pelz E, Erber R, Mohrmann S, Mobus V, Augustin D, Hoffmann G, Thomssen C, Janicke F, Kiechle M, Wallwiener D, Kuhn W, Nitz U, Harbeck N. Comparison of prognostic and predictive impact of genomic or central grade and immunohistochemical subtypes or IHC4 in HR+/HER2- early breast cancer: WSG-AGO EC-Doc Trial. Ann Oncol. 2016 Jun;27(6):1035-1040. doi: 10.1093/annonc/mdw070. Epub 2016 Feb 18. PMID 27022068